CLINICAL TRIAL: NCT03249129
Title: Identification of Autoantibodies and Autoantigens in the Cerebrospinal Fluid of Patients With Spinal Cord Trauma
Acronym: TRAME
Status: Withdrawn | Type: Observational
Why Stopped: sponsor decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_42; 2017-A00661-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-08-07; First posted 2017-08-15 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Bone Marrow Failure; Trauma
Keywords: Trauma; spinal cord; autoimmunity; antibody
MeSH Terms: conditions — Bone Marrow Failure Disorders; Wounds and Injuries; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to detect the presence of autoantibodies and autoantigens in cerebrospinal fluid early (<48 hours) following spinal cord trauma.

The study also aims to define the central or peripheral origin of autoantibodies by looking for their simultaneous presence at the blood level and to evaluate the prognostic value of the presence of autoantibodies within the cerebrospinal fluid, as well as on the initial clinical severity than on the recovery potential.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spinal cord injury dating back less than 48 hours
2. Men or women over 18 years of age
3. Patients benefiting from social protection
4. Surgery performed within 48 hours of the trauma
5. Informed and signed consent by the patient or trusted person

Exclusion Criteria:

1. Contra-indication to ensure surgical decompression within the first 48 hours following the trauma
2. Coagulation disorders or any condition that may make the lumbar puncture risky (eg, history of lumbar surgery)
3. Severe cranial trauma associated
4. History of autoimmune pathology
5. Immunosuppressive therapy or long-term corticosteroid therapy
6. Patients unable to comply with protocol requirements
7. Person benefiting from legal protection (guardianship / curator)
8. Person deprived of liberty
9. Patient unable to express consent
10. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years old with spinal cord trauma, for whom CSF sampling may be performed safely within the first 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Level of anti glial fibrillary acid protein antibodies | The sampling is performed at the initial stage, i.e. within 48 hours after trauma. The time between trauma and sampling is specified and measured in hours.
  Anti glial fibrillary acid protein antibodies measured into the cerebrospinal fluid

SECONDARY OUTCOMES:
Blood level of anti glial fibrillary acid protein antibodies | The sampling is performed at the initial stage, i.e. within 48 hours after trauma. The time between trauma and sampling is specified and measured in hours.
  Anti glial fibrillary acid protein antibodies measured into the blood
Severity of Neurological Impairment | in the initial phase, at day 7, at 1 months, 3 months, 6 months and 1 year
  Measured using the American Society Injury Association score

CONTACTS AND LOCATIONS:
Overall Officials: Fahed Zairi, MD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: No